CLINICAL TRIAL: NCT04455516
Title: Meniscus Repair With Simultaneous ACL Reconstruction: Clinical Outcomes，Failure Rates And Subsequent Processing
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2020024
Record Dates: First submitted 2020-06-25; First posted 2020-07-02 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: The ACL Rupture; Meniscus Injury
Keywords: meniscus; failure of repair; anterior cruciate ligament reconstruction; arthroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- repair group: The first operation in these patients was meniscus repair
  Interventions: Procedure: Meniscus repair; partial meniscectomy
- nonfailure group: These patients had a successful first operation
  Interventions: Procedure: Meniscus repair; partial meniscectomy
- failure group: In these patients, the first meniscus repair operation failed
  Interventions: Procedure: Meniscus repair; partial meniscectomy

INTERVENTIONS:
Procedure: Meniscus repair; partial meniscectomy — 69 cases of meniscus repair (repair group) and 96 cases of partial meniscectomy (partial meniscectomy group), were retrospectively analyzed. The 69 patients of the repair group were divided into the nonfailure group (62 cases) and the failure group (7 cases) depending on the repair effect.

SUMMARY:
Our study has explored the causes of failure of meniscus repair and investigated the clinical effects of partial meniscectomy when meniscus repair failed.

DETAILED DESCRIPTION:
Background: Meniscus repair performed during ACL reconstruction may fail and the subsequent treatment includes revision meniscal repair or partial meniscectomy.

Purpose: To retrospectively analyze the clinical outcomes of meniscus repair with simultaneous anterior cruciate ligament (ACL) reconstruction and explore the causes of failure of meniscus repair.

Methods: From May 2013 to July 2018, the clinical data of 165 patients who were treated with meniscus surgery and simultaneous ACL reconstruction by the same doctor, including 69 cases of meniscus repair (repair group) and 96 cases of partial meniscectomy (partial meniscectomy group), were retrospectively analyzed. The 69 patients of the repair group were divided into the nonfailure group (62 cases) and the failure group (7 cases) depending on the repair effect. The average follow-up period was 38 (±10.5) months. Postoperative outcomes of the repair group and the partial meniscectomy group were compared. General conditions and postoperative outcomes of the failure group and the nonfailure group were compared. Seven patients in the failure group who underwent second arthroscopy were followed up for 30 (±17.4) months, and their postoperative outcomes were summarized.

ELIGIBILITY:
Inclusion Criteria:

1. patients with intraoperatively confirmed ACL rupture combined with medial, lateral, or medial and lateral meniscal injury;
2. age <60 years
3. no history of previous ipsilateral knee meniscal injury.

Exclusion Criteria:

1. ACL rupture associated with fracture, collateral ligament injury, or complex ligament injury;
2. a history of knee surgery;
3. a significant degree of osteoarthritis.

Ages: 13 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This retrospective case series was conducted to evaluate the clinical outcomes and failure rates of primary meniscus repair with simultaneous ACL reconstruction in patients who were operated by the same physician at our institution.
Sampling Method: Non-Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2020-03-16 (Actual); Primary Completion 2020-04-16 (Actual); Study Completion 2020-05-16 (Actual)

PRIMARY OUTCOMES:
The result of partial meniscus resection | Two years after the surgery
  Clinical signs were assessed after the surgery, including swelling of the joint, tenderness at the joint line, locked-in syndrome, and positive McMurray's sign.
International Knee Documentation Committee（IKDC）scores | Two years after the surgery
  The minimum is 0, the maximum is 100, and the higher the score, the better the result
Visual analog scale (VAS) scores | Two years after the surgery
  The minimum is 0, the maximum is 10, and the higher the score, the worse the result
Lysholm scores | Two years after the surgery
  The minimum is 0, the maximum is 100, and the higher the score, the better the result

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No